CLINICAL TRIAL: NCT05193019
Title: Practice Patterns of Antithrombotic Therapy in REAL-world Patients Undergoing PCI in Spain: Parenteral Antiplatelet Agents
Brief Title: Parenteral Antiplatelet Agents in Real-world Spanish PCI Patients
Acronym: PATREAL
Status: Active, not recruiting | Type: Observational
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Other Study IDs: EPIC27-PATREAL
Record Dates: First submitted 2021-12-31; First posted 2022-01-14 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Ischemic Heart Disease; Acute Coronary Syndrome
Keywords: Percutaneous Coronary Intervention; Antiplatelet Drugs; Cangrelor; Glycoprotein IIb/IIIa inhibitors
MeSH Terms: conditions — Myocardial Ischemia; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing PCI
  Interventions: Other: Parenteral antiplatelet agents

INTERVENTIONS:
Other: Parenteral antiplatelet agents — Patients undergoing PCI and receiving parenteral antiplatelet agents, cangrelor or glycoprotein IIb/IIIa inhibitors (GPIs), during the procedure as per clinical practice

SUMMARY:
This registry will provide exploratory and descriptive information regarding contemporary practice patterns of parenteral antiplatelet therapy in the PCI (Percutaneous Coronary Intervention) setting and will investigate as well the short-term effectiveness and safety of the currently available parenteral antiplatelet agents in a cohort of "real-world" patients undergoing PCI in Spain.

DETAILED DESCRIPTION:
The present study is an observational, multicenter, nationwide, prospective investigation in patients undergoing PCI due to any coronary syndrome (acute or chronic) and receiving parenteral antiplatelet agents, GPIs or cangrelor, as per clinical practice during the procedure.

This investigation will provide exploratory and descriptive information regarding contemporary practice patterns of parenteral antiplatelet therapy in the PCI setting and will evaluate the short-term effectiveness and safety of the currently available parenteral antiplatelet agents in a cohort of patients undergoing PCI in Spain.

Approximately 15 high-volume PCI-capable Spanish centers will participate in the present investigation with the intention to enroll circa 1.000 patients.

The study is purely observational and no intervention will be performed in the included subjects because due to their participation in this investigation.

Patients fulfilling inclusion and exclusion criteria will be included after providing written informed consent to participate in the current investigation. Patient characteristics, procedural details and pharmacological therapies will be collected after inclusion and clinical events will be registered at two time points: 48 hours and 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Undergoing a PCI
* Use of a parenteral antiplatelet agent (GPIs or cangrelor)during the invasive procedure (PCI)

Exclusion Criteria:

* Blood dyscrasia, bleeding diathesis or active bleeding at the time of the index procedure.
* Chronic oral anticoagulation.
* Recent history of stroke, TIA (Transient Ischemic Attack)or intracranial bleeding (<3 months prior to inclusion).
* Severe anemia (Hb<9g/dl) or platelet count <100x106/ml at the time of the index procedure.
* Any active neoplasm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a PCI and use of a parenteral antiplatelet agent (GPIs or cangrelor)during the invasive procedure (PCI)
Sampling Method: Non-Probability Sample
Enrollment: 717 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Net Adverse Clinical Events (NACE) | 48 hours
  NACE defined as a the composite of all-cause death, recurrent myocardial infarction, stroke, target vessel revascularization, definite or probable stent thrombosis and BARC bleeding (type 2,3 and 5) will be evaluated at 48 hours from index procedure

SECONDARY OUTCOMES:
Death | 48 hours
  All-cause of death will be evaluated at 48 hours from index procedure
Myocardial infarction | 48 hours
  Recurrent myocardial infarction will be evaluated at 48 hours from index procedure
Stroke | 48 hours
  Stroke will be evaluated at 48 hours from index procedure
Target Vessel Revascularization | 48 hours
  Target Vessel will be evaluated at 48 hours from index procedure
Definite or probable stent thrombosis | 48 hours
  Definite or probable stent thrombosis will be evaluated at 48 hours from index procedure
BARC bleeding | 48 hours
  BARC bleeding (type 2,3 and 5) will be evaluated at 48 hours from index procedure
Rate of Net Adverse Clinical Events (NACE) | 30 days
  NACE defined as a the composite of all-cause death, recurrent myocardial infarction, stroke, target vessel revascularization, definite or probable stent thrombosis and BARC bleeding (type 2,3 and 5) will be evaluated at 30 days from index procedure
Death | 30 days
  All-cause of death will be evaluated at 30 days from index procedure
Myocardial infarction | 30 days
  Recurrent myocardial infarction will be evaluated at 30 days from index procedure
Stroke | 30 days
  Stroke will be evaluated at 30 days from index procedure
Target Vessel Revascularization | 30 days
  Target Vessel Revascularization will be evaluated at 30 days from index procedure
Definite or probable stent thrombosis | 30 days
  Definite or probable stent thrombosis will be evaluated at 30 days from index procedure
BARC bleeding | 30 days
  BARC bleeding will be evaluated at 30 days from index procedure
Cardiac death | 48 hours
  Cardiac death will be evaluated at 48 hours from index procedure
Cardiac death | 30 days
  Cardiac death will be evaluated at 30 days from index procedure
Transition to oral P2Y12 inhibitors | 24 hours
  Proportion of patients transitioned to each oral P2Y12 inhibitor (clopidogrel, prasugrel or ticagrelor) after the use of each parenteral antiplatelet agent (GPIs or cangrelor) will be evaluated at 24 hours from index procedure

CONTACTS AND LOCATIONS:
Locations (12):
- Spain (12):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario de Cruces, Barakaldo
  - Hospital de Galdakao, Galdakao
  - Hospital Universitario de Cabueñes, Gijón
  - H.de Leon, León
  - Hospital Central de La Defensa Gómez Ulla, Madrid
  - Hospital Universitario de Navarra, Pamplona
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Clinico Universitario Santiago de Compostela, Santiago de Compostela
  - Hospital Universitari Joan Xxiii, Tarragona
  - Hospital Universitario Lozano Blesa, Zaragoza

REFERENCES:
- [Background] Collet JP, Thiele H, Barbato E, Barthelemy O, Bauersachs J, Bhatt DL, Dendale P, Dorobantu M, Edvardsen T, Folliguet T, Gale CP, Gilard M, Jobs A, Juni P, Lambrinou E, Lewis BS, Mehilli J, Meliga E, Merkely B, Mueller C, Roffi M, Rutten FH, Sibbing D, Siontis GCM; ESC Scientific Document Group. 2020 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation. Eur Heart J. 2021 Apr 7;42(14):1289-1367. doi: 10.1093/eurheartj/ehaa575. No abstract available. PMID 32860058
- [Background] Capodanno D, Ferreiro JL, Angiolillo DJ. Antiplatelet therapy: new pharmacological agents and changing paradigms. J Thromb Haemost. 2013 Jun;11 Suppl 1:316-29. doi: 10.1111/jth.12219. PMID 23809135
- [Background] Bhatt DL, Stone GW, Mahaffey KW, Gibson CM, Steg PG, Hamm CW, Price MJ, Leonardi S, Gallup D, Bramucci E, Radke PW, Widimsky P, Tousek F, Tauth J, Spriggs D, McLaurin BT, Angiolillo DJ, Genereux P, Liu T, Prats J, Todd M, Skerjanec S, White HD, Harrington RA; CHAMPION PHOENIX Investigators. Effect of platelet inhibition with cangrelor during PCI on ischemic events. N Engl J Med. 2013 Apr 4;368(14):1303-13. doi: 10.1056/NEJMoa1300815. Epub 2013 Mar 10. PMID 23473369
- [Background] Steg PG, Bhatt DL, Hamm CW, Stone GW, Gibson CM, Mahaffey KW, Leonardi S, Liu T, Skerjanec S, Day JR, Iwaoka RS, Stuckey TD, Gogia HS, Gruberg L, French WJ, White HD, Harrington RA; CHAMPION Investigators. Effect of cangrelor on periprocedural outcomes in percutaneous coronary interventions: a pooled analysis of patient-level data. Lancet. 2013 Dec 14;382(9909):1981-92. doi: 10.1016/S0140-6736(13)61615-3. Epub 2013 Sep 3. PMID 24011551
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437